CLINICAL TRIAL: NCT04929210
Title: A Phase 4, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Bio-naive Participants With Active Psoriatic Arthritis Axial Disease
Brief Title: A Study of Guselkumab Administered Subcutaneously in Bio-naive Participants With Active Psoriatic Arthritis Axial Disease
Acronym: STAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109043; CNTO1959PSA4002 (Other: Janssen Research & Development, LLC); 2021-000465-32 (EudraCT Number); 2023-504716-15-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab and Placebo (Experimental): Participants will receive guselkumab and matching placebo subcutaneously (SC) to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab SC.
  Interventions: Drug: Guselkumab
- Group 3: Placebo followed by Guselkumab (Experimental): Participants will receive matching placebo and will cross over to receive guselkumab SC.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Other Names: TREMFYA
Drug: Placebo — Matching placebo will be administered as subcutaneous injection.
  Arms: Group 1: Guselkumab and Placebo; Group 3: Placebo followed by Guselkumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab treatment in participants with active psoriatic arthritis (PsA) axial disease by assessing reduction in axial symptoms and inflammation.

DETAILED DESCRIPTION:
PsA is a chronic inflammatory musculoskeletal disease that has 6 disease domains, and axial disease represents one of the domains. Guselkumab is a fully human immunoglobulin (Ig) G1 lambda monoclonal antibody (mAb) that by binding to the p19 protein subunit of interleukin (IL)-23, blocks the binding of extracellular IL-23 to the cell surface IL-23 receptor, inhibiting IL-23-mediated intracellular signaling, activation, and cytokine production. This study will consist of a screening phase (up to 6 weeks), a treatment phase (up to 48 weeks, including a placebo-controlled period from Week 0 to Week 24 and an active-controlled treatment phase from Week 24 to Week 48), and a safety follow-up phase (up to Week 60). The efficacy assessments will include assessment such as Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score and the safety assessments will include evaluations of physical examinations, vital signs, electrocardiograms, clinical laboratory tests, and adverse events. The overall duration of the study will be up to 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriatic arthritis (PsA) for at least 6 months prior to the first administration of study intervention and meet classification criteria for psoriatic arthritis (CASPAR) criteria at screening
* Have active PsA as defined by: a) at least 3 swollen joints and at least 3 tender joints at screening and at baseline and b) C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligram/deciliter (mg/dL) at screening from the central laboratory, and despite previous non-biologic disease modifying antirheumatic drug (DMARD), apremilast, and/or nonsteroidal anti-inflammatory drug (NSAID) therapy
* Have magnetic resonance imaging (MRI)-confirmed PsA axial disease (positive MRI spine and/or sacroiliac [SI] joints, shown by a Spondyloarthritis Research Consortium of Canada [SPARCC] score of >= 3 in either the spine or the sacroiliac joints)
* Have a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of at least 4, and have a spinal pain score (on a visual analog scale [VAS]) of at least 4
* Have active plaque psoriasis, with at least 1 psoriatic plaque of >= 2 centimeter (cm) diameter and/or nail changes consistent with psoriasis, or documented history of plaque psoriasis

Exclusion Criteria:

* Has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients
* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), ankylosing spondylitis (AS)/non-radiographic-axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, or Lyme disease
* Has previously received any biologic treatment
* Has ever received a Janus kinase (JAK) inhibitor including but not limited to tofacitinib, baricitinib, filgotinib, peficitinib, decernotinib, upadacitinib or any other investigational JAK inhibitor
* Has received any systemic immunosuppressants (example, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2027-04-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Week 24 | Baseline and Week 24
  BASDAI is a self-assessment tool that consists of 6 questions relating to 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain, enthesitis, qualitative morning stiffness and quantitative morning stiffness. First 5 items were scored on a 10 centimeter (cm) visual analog scale (VAS) ranging from 0 equals to (=) none to 10=very severe. Quantitative morning stiffness was scored on a 10 cm VAS ranging from 0=0 hours to 10=2 or more hours. 2 scores for qualitative and quantitative morning stiffness were averaged, and total BASDAI score was average of the 5 scores of each symptom, ranging from 0 (none) to 10 (very severe). Higher scores indicate greater disease severity.

SECONDARY OUTCOMES:
Change from Baseline in Ankylosing Spondylitis Disease Activity Score-C-Reactive Protein (ASDAS-CRP) at Week 24 | Baseline and Week 24
  The ASDAS-CRP is a composite of 5 disease activity variables with only partial overlap. The 4 self-reported items included in this index are back pain (VAS), duration of morning stiffness, peripheral pain/swelling, and participant global assessment of disease activity; these are combined with the C-reactive protein (CRP) value. Selected cut-offs for improvement scores are: a change greater than or equal to (>=) 1.1 units for "clinically important improvement" and a change >= 2.0 units for "major improvement.
Change from Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) at Week 24 | Baseline and Week 24
  DAPSA assessed the joint domain of psoriatic arthritis (PsA) and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (milligram/deciliter [mg/dL], value less than [<] lower limit of quantification [LLOQ] is considered equal to half of the value of LLOQ for numerical calculations), participant assessment of pain (0-10 cm VAS, 0=no pain, 10=worst possible pain), and participant's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. The assessment does not have a score range with an upper or lower bound.
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 24 | Baseline and Week 24
  HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Percentage of Participants with Investigator's Global Assessment (IGA) 0/1 Response at Week 24 among Participants with >= 3% Body Surface Area (BSA) Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline | Week 24
  Percentage of participants with IGA 0/1 response at week 24 among the participants with >= 3 percent (%) BSA psoriatic involvement and an IGA score of >= 2 (mild) at baseline will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given timepoint. Overall lesions are graded for induration, erythema, and scaling using 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate) and 4 (severe) scale. The IGA score of psoriasis is based upon the average of induration, erythema and scaling scores. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Change from Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Score for Magnetic Resonance Imaging (MRI) Sacroiliac (SI) Joints at Week 24 | Baseline and Week 24
  Change from baseline in SPARCC score for MRI SI joints at week 24 among the participants with a positive MRI of the sacroiliac joints at baseline will be reported. SPARCC method focuses on the cartilaginous portion of the SI joint, and scores presence (score of 1) versus absence (score of 0) of bone marrow edema in each SI joint quadrant.
Percentage of Participants who Achieve a >= 50 % Improvement from Baseline in BASDAI Score at Week 24 | Baseline and Week 24
  Percentage of participants who achieve a >= 50 % improvement from baseline in BASDAI score at week 24 will be reported.
Percentage of Participants who Achieve ASDAS Clinically Important Improvement at Week 24 | Week 24
  Percentage of participants who achieve ASDAS clinically important improvement at week 24 will be reported.
Percentage of Participants who Achieve Ankylosing Spondylitis Activity Score (ASAS) 40 Response at Week 24 | Week 24
  Percentage of participants who achieve ASAS 40 response at Week 24 will be reported. ASAS 40 defined as improvement from baseline of >= 40% and with an absolute improvement from baseline of at least 2 on 0 to 10 cm scale in at least 3 of following 4 domains: Participant's global assessment (0 to 10 cm; 0=very well, 10=very poor), total back pain (0 to 10 cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10 cm; 0=none, 10=very severe); no worsening at all from baseline in remaining domain.
Percentage of Participants who Achieve ASDAS Major Improvement at Week 24 | Week 24
  Percentage of participants who achieve ASDAS major improvement at Week 24 will be reported.
Change from Baseline in SPARCC Score for MRI Spine at Week 24 | Baseline and Week 24
  Change from baseline in SPARCC score for MRI spine at week 24 among the participants with a positive MRI of the spine at baseline will be reported. The SPARCC scoring system for the spine scores the 6 discovertebral units considered by the reader as the most abnormal, and then separately assesses each quadrant of 3 adjacent sagittal slices, with additional points for "depth" and high "intensity" of the lesion.
Number of Participants with Adverse Events (AEs) | Up to 60 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious Adverse Events (SAEs) | Up to 60 weeks
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Reasonably Related AEs | Up to 60 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs Leading to Discontinuation of Study Intervention | Up to 60 weeks
  Number of participants with AEs leading to discontinuation of study intervention will be reported.
Number of Participants with Infections | Up to 60 weeks
  Number of participants with infections will be reported.
Number of participants with Injection-Site Reactions | Up to 60 weeks
  Number of participants with injection-site reactions will be reported. A study intervention injection-site reaction is any adverse reaction at a subcutaneous study intervention injection-site.
Number of Participants with Laboratory Abnormalities (Chemistry, Hematology) by Maximum Toxicity (Common Terminology Criteria for Adverse Events [CTCAE 5.0]) Grades | Up to 60 weeks
  Number of participants with laboratory abnormalities (chemistry, hematology) by maximum toxicity (CTCAE 5.0) grades will be reported. Grade refers to the severity of the AE as follows: Grade 1- Mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2- Moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental Activities of Daily Living (ADL); Grade 3- Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self-care ADL; Grade 4- Life-threatening consequences, urgent intervention indicated; Grade 5- Death related to AE.
Serum Guselkumab Concentration Over Time | Up to 60 weeks
  Serum guselkumab concentration over time will be reported.
Number of Participants with Antibodies to Guselkumab | Up to 60 weeks
  Number of participants with antibodies to guselkumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (240):
- United States (38):
  - Arizona Arthritis and Rheumatology Research PLLC, Avondale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Chandler, Arizona
  - Arizona Arthritis and Rheumatology Research PLLC, Mesa, Arizona
  - Arizona Arthritis Research, PLC., Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Associates, Sun City, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - Unity Health-White County Medical Center, Searcy, Arkansas
  - Kaiser Permanent Medical Center, Fontana, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - University Of California San Diego, La Jolla, California
  - Rheumatology Center of San Diego, San Diego, California
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - OrthoIllinois, Rockford, Illinois
  - Willow Rheumatology and Wellness, Willowbrook, Illinois
  - Johns Hopkins Bayview Medical, Baltimore, Maryland
  - Klein And Associates M D P A, Hagerstown, Maryland
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology P A, Eagan, Minnesota
  - Kansas City Physician Partners, Kansas City, Missouri
  - Clinvest, Springfield, Missouri
  - STAT Research, Inc., Vandalia, Ohio
  - OHSU Rheumatology Clinic, Marquam Hill, Portland, Oregon
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Adriana Pop Moody MD Clinic PA, Corpus Christi, Texas
  - AARA Clinical Research Lone Star Arthritis and Rheumatology, Fort Worth, Texas
  - UT Physicians Center for Autoimmunity, Houston, Texas
  - AARA Clinical Research Lone Star Arthritis and Rheumatology, Irving, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Epic Medical Research, Red Oak, Texas
  - DM Clinical Research, Tomball, Texas
  - Swedish Medical Center, Seattle, Washington
- Argentina (6):
  - Cosultorios Reumatologógicos Pampa, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Hospital Italiano La Plata, La Plata
  - MR Medicina Reumatologica, San Fernando
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Australia (6):
  - Emeritus Research, Camberwell
  - Southern Clinical Research, Hobart
  - Liverpool Hospital, Liverpool
  - Rheumatology Research Unit, Maroochydore
  - Skin Health Institute Inc., Melbourne
  - Eastern Health - Box Hill Hospital, Melbourne
- Bulgaria (13):
  - Exacta Medica, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Medical Center Unimed Plovdiv, Plovdiv
  - UMHAT Kaspela, Plovdiv
  - Medical Center Artmed, Plovdiv
  - MHAT 'Lyulin' EAD, Sofia
  - University Multiprofile Hospital Sofiamed Sofia, Sofia
  - Military Medical Academy, Sofia
  - UMHAT St. Ivan Rilski, Sofia
  - DCC Convex EOOD, Sofia
  - ASIMP Rheumatology Centre St Irina EOOD, Sofia
  - Medical Centre Synexus, Sofia
  - DDC Sv. Ivan Rilski OOD, Targovishte
- Canada (4):
  - Skin Care Centre, Vancouver, British Columbia
  - Eastern Regional Health Authority St Clares Mercy Hospital, St. John's, Newfoundland and Labrador
  - Toronto Western Hospital, Toronto, Ontario
  - G R M O Groupe de recherche en maladies osseuses Inc, Québec, Quebec
- Czechia (9):
  - Revmaclinic, Brno
  - Revmatologie s r o, Brno
  - Revmacentrum MUDr Mostera s r o, Brno-Židenice
  - L K N Arthrocentrum, Hlučín
  - Revimex Pro s r o, Karvina Frystat
  - MUDr Rosypalova s r o, Ostrava
  - Arthrohelp S.R.O., Pardubice
  - Revmatologicky ustav, Prague
  - Medical Plus S R O, Uherské Hradiště
- Denmark (4):
  - Frederiksberg Hospital, Frederiksberg
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Køge Sygehus Region Sjaelland, Køge
  - Vejle Sygehus, Vejle
- Georgia (15):
  - Ltd Health Center, Batumi
  - LTD Clinic LJ, Kutaisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - Ltd American Hospital Network, Tbilisi
  - LTD Helsicore, Tbilisi
  - Ltd New Hospitals, Tbilisi
  - TSMU The First University Clinic, Tbilisi
  - JSC K Eristavi National Center of experimental and Clinical surgery, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd, Tbilisi
  - LTD 'Aversi Clinic', Tbilisi
  - LTD MediClub Georgia, Tbilisi
  - Clinic on Mtskheta Street, Tbilisi
  - LTD The First Medical Center, Tbilisi
  - Consilium Medulla-multiprofile clinic Ltd, Tbilisi
  - JSC Evex Hospitals, Tnilisi
- Germany (4):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumazentrum Ratingen, Ratingen
- Prince Of Wales Hospital, Hong Kong, Hong Kong
- Hungary (8):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Qualiclinic Kft, Budapest
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Porcika Klinika - Vasarhelyi Sarkanyfu Kft., Hódmezővásárhely
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Italy (6):
  - A.O. Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero-Universitaria di Cagliari, Monserrato
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Policlinico Tor Vergata, Roma
  - Humanitas Hospital, Rozzano (MI)
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Malaysia (5):
  - Hospital Selayang, Batu Caves
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tuanku Jaafar, Seremban
- Philippines (7):
  - Cebu Doctors' University Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - Lipa Medix Medical Hospital, Lipa
  - ManilaMed Medical Center Manila, Manila
  - Philippine General Hospital, Manila
  - St. Luke's Medical Center, Quezon City
  - Ilocos Training and Regional Medical Center, San Fernando City
- Poland (26):
  - ClinicMed Daniluk Nowak Spolka Komandytowa, Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela, Bydgoszcz
  - Nzoz Bif Med, Bytom
  - Ambulatorium sp. z o.o., Elblag
  - Centrum Kliniczno Badawcze, Elblag
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Centrum Medyczne Promed, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Centrum Medyczne AMED oddzial w Lodzi, Lodz
  - Velocity Lublin, Lublin
  - Reumed Zespol Poradni Specjalistycznych Filia nr 1, Lublin
  - Pro Life Medica Sp. z o.o., Lublin
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Twoja Przychodnia PCM, Poznan
  - Reumedika s c Wieslawa Porawska Lukasz Porawski, Poznan
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - MICS Centrum Medyczne Torun, Torun
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Rheuma Medicus Sp z o o, Warsaw
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - ETG Warszawa, Warsaw
  - Centrum Medyczne AMED Targowek, Warsaw
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Portugal (8):
  - Uls Braga - Hosp. Braga, Braga
  - Ulsg - Hosp. Sousa Martins, Guarda
  - Ipr Inst Port de Reumatologia, Lisbon
  - Uls Lisboa Ocidental - Hosp. Egas Moniz, Lisbon
  - Hosp. Cuf Tejo, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Ulsam - Hosp. Conde de Bertiandos, Ponte de Lima
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- Russia (21):
  - Altay Medical State University, Barnaul
  - Chelyabinck Regional Clinical Hospital, Chelyabinsk
  - Chelyabinsk Regional Clinical Dermatovenerological Dispensary, Chelyabinsk
  - Regional Clinical Diagnostic Center of Udmurtia Region, Izhevsk
  - LLL Medical Center Revma-Med, Kemerovo
  - LLC Family Outpatient Clinic # 4, Korolyov
  - Regional SBI of PH Krasnoyarsk Regional Clinical hospital #20 named after I.S. Berzon, Krasnoyarsk
  - Clinical-Diagnostic Center Euromedservice, JSC, Moscow
  - FGBU Research Institute of Rheumatology named V.A.Nasonova, Moscow
  - GBUZ of Moscow Region 'Moscow Region SRI n.a. Vladimirskyi', Moscow
  - Llc Ultramed, Omsk
  - GBOU VPO Orenburg State Medical University, Orenburg
  - GBUZ Perm Regional Clinical Hospital, Perm
  - Republican Hospital n.a.V.A.Baranov, Petrozavodsk
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - St. Petersburg GBUZ Clinical Reumatological Hospital 25, Saint Petersburg
  - X7 Clinical Research Company Limited, Saint Petersburg
  - GBUZ of Samara Region 'Tolyatti City Clinical Hospital 5', Tolyatti
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
  - Clinical Hospital #3, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital N. 1, Yekaterinburg
- Slovakia (5):
  - Reumatologicka ambulancia, Martin
  - Reumatologicka ambulancia, Nové Mesto nad Váhom
  - Reumatologická ambulancia Thermium s.r.o., Piešťany
  - REUMAMED POPRAD, s.r.o., Poprad
  - Reumex s.r.o, Rimavská Sobota
- Spain (12):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Hosp. Clinico San Carlos, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Clinica Gaias, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Quiron Sagrado Corazon, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset, Solna
  - Akademiska Sjukhuset, Uppsala
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Chiang Mai University, Chiang Mai
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Uludag University Medical Faculty, Bursa
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- Ukraine (13):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Municipal non-commercial enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - City Clinical Hospital No. 2, Kryvyi Rih
  - Medical Center of 'Institute of Rheumatology', LLC, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil
  - Health Clinic Limited Liability Company, Vinnytsia
  - Medical Center LLC 'Modern Clinic', Zaporizhzhya
- United Kingdom (7):
  - Royal Free London NHS Foundation Trust, Barnet
  - St. Lukes Hospital, Bradford
  - University Hospital Coventry & Warwickshire NHS Trust, Coventry
  - Chapel Allerton Hospital, Leeds
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - North Tyneside General Hospital, Newcastle
  - Haywood Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gladman DD, Mease PJ, Bird P, Soriano ER, Chakravarty SD, Shawi M, Xu S, Quinn ST, Gong C, Leibowitz E, Poddubnyy D, Tam LS, Helliwell PS, Kavanaugh A, Deodhar A, Ostergaard M, Baraliakos X. Efficacy and safety of guselkumab in biologic-naive patients with active axial psoriatic arthritis: study protocol for STAR, a phase 4, randomized, double-blinded, placebo-controlled trial. Trials. 2022 Sep 5;23(1):743. doi: 10.1186/s13063-022-06589-y. PMID 36064592